CLINICAL TRIAL: NCT05440838
Title: Identification of Factors Associated With Treatment Response in Patients With Polycythemia Vera, Essential Thrombocythemia, and Pre-myelofibrosis.
Acronym: BioPredictor
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: University Hospital, Brest (Other); Nantes University Hospital (Other); Poitiers University Hospital (Other); Rennes University Hospital (Other); University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01044-39
Record Dates: First submitted 2022-06-10; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Next-generation sequencing — Next-generation sequencing and cytokine profile will be established in all patients before the start of treatment.
  Other Names: Cytokines

SUMMARY:
First-line treatment for patients with polycythemia vera, essential thrombocythemia, and pre-myelofibrosis is based on hydroxyurea or pegylated interferon. The objective of treatment is to prevent thrombotic complications and leukemic transformation. Despite overall good response rates, some patients do not respond to treatment and others lose their response over time. Both situations are associated with worse survival and there are to date no clear predictive factors for response although the existence of additional mutations seems unfavorable.

In this exploratory study, we hypothesize that biological factors at diagnosis are associated with hematological response at 12 months. We will more specifically study the association between mutational profile, assessed by next-generation sequencing, and cytokine profile with hematological response.

This study will help in identifying patients who will not respond to hydroxyurea or pegylated interferon and give the opportunity to try other treatments upfront, in the perspective of precision medicine. On the basic science side, this study will help in understanding the molecular and immunological factors involved in resistance to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with polycythemia vera, essential thrombocythemia, or pre-myelofibrosis.
* Indication for first-line treatment with hydroxyurea or pegylated interferon.
* Consent to participate.
* Affiliated to social security.

Exclusion Criteria:

* Previous treatment.
* Other on-going malignancy, including overt myelofibrosis.
* Other treatment such as phlebotomy solely, ruxolitinib, anagrelide, or pipobroman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with polycythemia vera, essential thrombocythemia, or pre-myelofibrosis requiring first-line treatment with hydroxyurea or pegylated interferon.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-09-08 (Estimated); Primary Completion 2024-09-07 (Estimated); Study Completion 2029-10-04 (Estimated)

PRIMARY OUTCOMES:
Complete hematological response | 12 months
  ELN-2013 criteria by meeting all of the following:
  * Durable resolution of disease-related signs including palpable hepatosplenomegaly, large symptoms improvement, AND
  * Durable peripheral blood count remission, defined as: platelet count ≤400 ×109/L, WBC count <10 × 109/L, Ht lower than 45% without phlebotomies (for PV patients), absence of leukoerythroblastosis, AND
  * Without signs of progressive disease, and absence of any hemorrhagic or thrombotic events.

SECONDARY OUTCOMES:
Complete hematological response | 24, 36, 48, and 60 months
  ELN-2013 criteria by meeting all of the following:
  * Durable resolution of disease-related signs including palpable hepatosplenomegaly, large symptoms improvement, AND
  * Durable peripheral blood count remission, defined as: platelet count ≤400 ×109/L, WBC count <10 × 109/L, Ht lower than 45% without phlebotomies (for PV patients), absence of leukoerythroblastosis, AND
  * Without signs of progressive disease, and absence of any hemorrhagic or thrombotic events.
Molecular response | 12 and 24 months
  ELN-2013 criteria: Complete response is defined as eradication of a preexisting abnormality (CALR, JAK2, or MPL mutations) by quantitative PCR. Partial response applies only to patients with at least 20% mutant allele burden at baseline. Partial response is defined as ≥50% decrease in allele burden by quantitative PCR.

IPD SHARING:
Plan to Share IPD: Undecided